CLINICAL TRIAL: NCT00155376
Title: Intravenous-Morphine and Glucagon-Usage Enhanced MR Cholangiography
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 940104
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2005-11-28 (Estimated); Status verified 2005-04

CONDITIONS: Liver Disease
MeSH Terms: conditions — Liver Diseases | interventions — Morphine; Glucagon

INTERVENTIONS:
Drug: morphine and glucagon

SUMMARY:
Morphine can induce constriction of sphincter of oddi and glucagon can facilitate bile secretion and dilatation of bile duct. We conduct this randomized double blinded study to evaluate the effect of enhancement in MRCP using intravenous morphine and glucagon.

DETAILED DESCRIPTION:
Morphine can induce constriction of sphincter of oddi and glucagon can facilitate bile secretion and dilatation of bile duct. We conduct this randomized double blinded study to evaluate the effect of enhancement in MRCP using intravenous morphine and glucagon.

ELIGIBILITY:
Inclusion Criteria:

* normal volunteer
* living liver donor

Exclusion Criteria:

* COPD
* chronic liver disease
* hypersensitive to glucagon
* DM
* insulinoma
* glucagonoma
* pregnancy

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2005-09; Study Completion 2005-09

PRIMARY OUTCOMES:
MRCP visibility

CONTACTS AND LOCATIONS:
Overall Officials: Hon-Man Liu, MD, Study Chair — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Province of Taiwan, Taiwan